CLINICAL TRIAL: NCT00104689
Title: Phase II Trial Assessing the Impact on the Activity of Daily Living of an Oral Chemotherapy by Capecitabine Associated With an Intravenous Chemotherapy by Oxaliplatin as First Line Treatment of Metastatic Colorectal Adenocarcinoma of Patients Aged Over 70
Brief Title: Capecitabine and Oxaliplatin in Treating Older Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000416120; FRE-FNCLCC-GERICO-02/0301; EU-20500
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capecitabine + Oxaliplatin (Experimental): Patients receive oral capecitabine once daily on days 1-14 and oxaliplatin IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well giving capecitabine together with oxaliplatin works in treating older patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of capecitabine and oxaliplatin as first-line treatment, as defined by stabilization or improvement by 1 point on Katz's Activities of Daily Living scale, in older patients with metastatic colorectal adenocarcinoma.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the percentage of patients who receive the first 3 courses of this regimen (at lower doses) and the percentage of patients who receive all 6 courses of this regimen (at both lower and higher doses).
* Determine efficacy of this regimen, as defined by RECIST criteria, in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter, open-label, nonrandomized study.

Patients receive oral capecitabine* once daily on days 1-14 and oxaliplatin* IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *The doses of both capecitabine and oxaliplatin are increased in courses 4-6 in the absence of unacceptable toxicity

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal adenocarcinoma

  * Metastatic disease
* Requires first-line therapy for metastatic disease

PATIENT CHARACTERISTICS:

Age

* Over 70

Performance status

* Katz's Activities of Daily Living scale < 6 (≤ 6 for patients ≥ 80 years of age)

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* AST and ALT < 2 times normal (5 times normal if due to hepatic metastases)
* Bilirubin < 2 times normal (5 times normal if due to hepatic metastases)

Renal

* Creatinine clearance > 30 mL/min

Other

* No clinical neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 6 months since prior adjuvant chemotherapy
* No prior chemotherapy for metastatic disease

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-06-30 (Actual); Primary Completion 2007-03-31 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of stabilization or improvement by 1 point on Katz's Activities of Daily Living scale

SECONDARY OUTCOMES:
Toxicity
Percentage of patients who receive the first 3 treatment courses at a lower dose and the percentage of patients who receive all 6 treatment courses at both lower and higher doses
Efficacy as defined in RECIST criteria
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Viret, MD — Institut Paoli-Calmettes
Locations (9):
- France (9):
  - Centre Regional Francois Baclesse, Caen
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Polyclinique Francheville, Périgueux
  - Institut Jean Godinot, Reims
  - Centre Rene Huguenin, Saint-Cloud
  - C.H. Senlis, Senlis
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Viret F, Bugat R, Ducreux M, et al.: XELOX regimen in elderly patients with metastatic colorectal cancer (MCRC), a FNCLCC French Collaborative Group GERICO 02 phase II study. [Abstract] J Clin Oncol 25 (Suppl 18): A-19513, 708s, 2007.